CLINICAL TRIAL: NCT07241936
Title: A Phase Ib/II Clinical Trial on the Safety and Efficacy of Sirolimus (Albumin-bound) Combined With Different ADCs in Patients With Advanced Solid Tumors
Brief Title: A Study of Sirolimus (Albumin-Bound) in Combination With Different ADCs Treatment of Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HB1901-012
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Intervention Model Description: Dose escalation and expansion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- sirolimus (albumin-bound)+ DP303c (Experimental)
  Interventions: Drug: sirolimus (albumin-bound); Drug: DP303c
- sirolimus (albumin-bound)+ SYS6043 (Experimental)
  Interventions: Drug: sirolimus (albumin-bound); Drug: SYS6043
- sirolimus (albumin-bound)+ SYS6002 (Experimental)
  Interventions: Drug: sirolimus (albumin-bound); Drug: SYS6002
- sirolimus (albumin-bound)+ SYS6010 (Experimental)
  Interventions: Drug: sirolimus (albumin-bound); Drug: SYS6010

INTERVENTIONS:
Drug: sirolimus (albumin-bound) — intravenous infusion
Drug: DP303c — intravenous infusion
  Arms: sirolimus (albumin-bound)+ DP303c
Drug: SYS6043 — intravenous infusion
  Arms: sirolimus (albumin-bound)+ SYS6043
Drug: SYS6002 — intravenous infusion
  Arms: sirolimus (albumin-bound)+ SYS6002
Drug: SYS6010 — intravenous infusion
  Arms: sirolimus (albumin-bound)+ SYS6010

SUMMARY:
This study adopts a multi-center, open-label, non-randomized trial design. It plans to enroll patients with Advanced solid tumor. Dose-escalation and PK-expansion studies will be carried out to evaluate the safety, tolerability, and preliminary efficacy of sirolimus (albumin-bound) in combination with Different ADCs (DP303c/SYS6043/SYS6002/SYS6010) in this patient population, and to confirm the recommended phase 2 dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects aged 18 to 75 years (inclusive).
* 2. Patients with advanced solid tumors that are unresectable or metastatic and confirmed by histology or cytology.
* 3. At least one measurable lesion, as defined by RECIST 1.1 criteria.
* 4. ECOG performance status of 0 or 1.
* 5. Expected survival ≥ 3 months.
* 6. Adequate function of major organs and bone marrow.
* 7. Willing to provide samples of previously removed tumors or undergo fresh tumor biopsy.
* 8. Women or man of childbearing potential must use highly effective contraception.
* 9. Able to understand and voluntarily sign the written informed consent form (ICF).

Exclusion Criteria:

* 1. Previous use of antibody-conjugated drugs with similar loading agents for treatment.
* 2. Previous anti-tumor treatment drugs were not adequately removed.
* 3. Active leptomeningeal disease or uncontrolled CNS metastasis.
* 4. Having a history of severe or uncontrolled cardiovascular or cerebrovascular diseases.
* 5. Previous interstitial lung disease requiring glucocorticoid treatment, Or currently suffering from interstitial lung disease/non-infectious pneumonia, or the imaging examination during the screening period cannot rule out interstitial pneumonia/lung disease.
* 6. Patients who developed severe and moderately severe lung diseases that significantly affected lung function within 6 months of the first medication administration; patients requiring supplementary oxygen therapy.
* 7. Individuals who currently have eye diseases such as corneal disorders, retinal disorders, or active ocular infections that require intervention, or who have a history of serious corneal-related eye diseases in the past; or who are unwilling to stop wearing corneal contact lenses during the study; or who have other existing eye diseases that affect the assessment of ocular toxicity after the administration of the investigational drug.
* 8. Currently suffering from skin diseases that require oral or intravenous medication treatment.
* 9. Had a history of ulcerative colitis or Crohn's disease.
* 10. Within 14 days prior to the first administration of the medication, there is a need for systemic antibacterial, antifungal or antiviral treatment for severe chronic or active infections, and there is no cure for active tuberculosis.
* 11. Known to be allergic to any component of the test drug, or allergic to the humanized monoclonal antibody product.
* 12. Participants with poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
The occurrence and frequency of adverse events (AE) and serious adverse events (SAE) | Up to approximately 36 weeks after the first participant is enrolled
dose - limiting toxicities (DLT) | Up to approximately 36 weeks after the first participant is enrolled
The recommended phase 2 dose | Up to approximately 36 weeks after the first participant is enrolled

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China